CLINICAL TRIAL: NCT02173639
Title: Relative Oral Bioavailability of a Fixed Dose Combination Tablet of BI 1356 2.5 mg / Metformin 1000 mg, Compared With Single BI 1356 2.5 mg and Metformin 1000 mg Tablets Administered Together to Healthy Male and Female Subjects in an Open, Randomised, Single-dose, Two-way Crossover, Phase I Trial
Brief Title: Bioavailability of Combination Tablet BI 1356/Metformin Compared With Single BI 1356 and Metformin Administered Together to Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.47
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (2):
- BI 1356/metformin (Experimental)
  Interventions: Drug: BI 1356/metformin
- BI 1356 + Metformin (Experimental)
  Interventions: Drug: BI 1356; Drug: Metformin

INTERVENTIONS:
Drug: BI 1356/metformin — fixed dose combination tablet
  Arms: BI 1356/metformin
Drug: BI 1356
  Arms: BI 1356 + Metformin
Drug: Metformin
  Arms: BI 1356 + Metformin

SUMMARY:
The objective was to assess the relative bioavailability of a pilot scale linagliptin 2.5 mg / metformin 1000 mg fixed dose combination (FDC) tablet in comparison with single tablets of linagliptin 2.5 mg and metformin 1000 mg administered together.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females based upon a complete medical history, including the physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead Electrocardiogram, clinical laboratory tests
* Age ≥18 and ≤ 55 years
* BMI ≥18.5 and ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination deviating from normal and of clinical relevance. Repeated measurement of a systolic blood pressure greater than 140 mm Hg or a diastolic blood pressure greater than 90 mm Hg
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration and during the trial except if a relevant interaction can be ruled out
* Participation in another trial with an investigational drug within two months prior to first study drug administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on pharmacokinetic study days
* Alcohol abuse (average consumption of more than 20 g/day in females and more than 30 g/day in males)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to the start of study)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 450 ms)
* A history of additional risk factors for Torsade de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For female subjects:

* Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion
* No adequate contraception during the study and until 2 months after study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, IUD (intrauterine device), sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to use an additional barrier method (e.g. condom, diaphragm with spermicide)
* Lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
AUC0-72 h (area under the concentration-time curve of BI 1356 in plasma over the time interval from 0 to 72 h) | up to 72 hours after administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 168 hours after administration
AUC0-∞ (area under the concentration-time curve of metformin in plasma over the time interval from 0 to infinity) | up to 168 h after administration

SECONDARY OUTCOMES:
tmax (time from dosing to maximum concentration of the analyte in plasma) | up to 168 hours after administration
λz (terminal elimination rate constant of the analyte in plasma) | up to 168 hours after administration
t1/2 (terminal half-life of the analyte in plasma) | up to 168 hours after administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 168 hours after administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 168 hours after administration
Vz/F (apparent volume of distribution during the terminal phase λz of the analyte following an extravascular dose) | up to 168 hours after administration
Number of patients with adverse events | up to 11 weeks
Assessment of tolerability on a 4-point scale by investigator | 14 days after last study drug administration
AUC0-24 h (area under the concentration-time curve of BI 1356 and metformin in plasma over the time interval from 0 to the 24 h) | up to 24 h after administration
AUC0-tz (area under the concentration-time curve of BI 1356 and metformin in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 168 h after administration
AUC0-∞ (area under the concentration time curve of BI 1356 in plasma over the time interval from 0 extrapolated to infinity) | up to 168 h after administration